CLINICAL TRIAL: NCT01294462
Title: A Randomised, Double-blind, Double-dummy, Parallel Group, International (Asian), Multicenter, Phase 3 Study to Assess Safety and Efficacy of AZD6140 on Top of Low Dose Acetyl Salicylic Acid (ASA) Versus Clopidogrel on Top of Low Dose ASA in Asian/Japanese Patients With Non-ST or ST Elevation Acute Coronary Syndromes(ACS) for Whom PCI is Planned
Brief Title: Study to Assess Safety and Efficacy of Ticagrelor (AZD6140) Versus Clopidogrel in Asian/Japanese Patients With Non-ST or ST Elevation Acute Coronary Syndromes (ACS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5130C00027
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Acute Coronary Syndrome; Percutaneous Coronary Intervention
Keywords: acute coronary syndrome; coronary disease; coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Disease; Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Ticagrelor (AZD6140)
  Interventions: Drug: Ticagrelor; Drug: Acetylsalicylic acid ASA
- 2 (Active Comparator): Clopidogrel
  Interventions: Drug: Clopidogrel; Drug: Acetylsalicylic acid ASA

INTERVENTIONS:
Drug: Ticagrelor — 90 mg, oral dose twice daily
  Other Names: AZD6140
  Arms: 1
Drug: Clopidogrel — 75 mg, oral dose once daily
  Other Names: Plavix
  Arms: 2
Drug: Acetylsalicylic acid ASA — Low Dose ASA

SUMMARY:
The purpose of the study is to assess the efficacy (prevention of vascular events) and safety (especially bleedings) of Ticagrelor (AZD6140) compared with Clopidogrel, both given on top of low dose aspirin, in Asian/Japanese patients with acute coronary syndrome and a planned percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent
* Index event of non-ST or ST segment elevation ACS

Exclusion Criteria:

* Index event is an acute complication of percutaneous coronary intervention
* Patient has undergone Percutaneous Coronary Intervention (PCI) after the index event before the first dose of study treatment
* Oral anticoagulation therapy that cannot be stopped
* The conditions associated with increased risk of bradycardiac events

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hsia, MD, Study Director — AstraZeneca
Locations (87):
- Japan (79):
  - Research Site, Ichinomiya-shi, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Okazaki-shi, Aichi-ken
  - Research Site, Toyohashi, Aichi-ken
  - Research Site, Toyota-shi, Aichi-ken
  - Research Site, Akita, Akita
  - Research Site, Ichihara-shi, Chiba
  - Research Site, Kamogawa-shi, Chiba
  - Research Site, Kisarazu-shi, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukui-shi, Fukui
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kasuya-gun, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Gifu, Gifu
  - Research Site, Isesaki, Gunma
  - Research Site, Maebashi, Gunma
  - Research Site, Takasaki-shi, Gunma
  - Research Site, Kure, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Akashi-shi, Hyōgo
  - Research Site, Amagasaki-shi, Hyōgo
  - Research Site, Kawanishi-shi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Nishinomiya, Hyōgo
  - Research Site, Takarazuka-shi, Hyōgo
  - Research Site, Higashiibaragi-gun, Ibaragi
  - Research Site, Sashima-gun, Ibaragi
  - Research Site, Hakusan-shi, Ishikawa-ken
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Sakaide-shi, Kagawa-ken
  - Research Site, Atsugi-shi, Kanagawa
  - Research Site, Isehara, Kanagawa
  - Research Site, Kamakura-shi, Kanagawa
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Yamato-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Nankoku-shi, Kochi
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Yatsushiro, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Azumino-shi, Nagano
  - Research Site, Ueda-shi, Nagano
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Ōita, Oita Prefecture
  - Research Site, Kurashiki, Okayama-ken
  - Research Site, Okayama, Okayama-ken
  - Research Site, Hirakata, Osaka
  - Research Site, Kawachinagano-shi, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Sakai-shi, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Ageo-shi, Saitama
  - Research Site, Hidaka, Saitama
  - Research Site, Sayama-shi, Saitama
  - Research Site, Kusatsu-shi, Shiga
  - Research Site, Moriyama, Shiga
  - Research Site, Matsue, Shimane
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Izunokuni, Shizuoka
  - Research Site, Shimada-shi, Shizuoka
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Komatsushima-shi, Tokushima
  - Research Site, Tokushima, Tokushima
  - Research Site, Adachi-ku, Tokyo
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Bunkyo, Tokyo
  - Research Site, Chiyoda-ku, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Meguro City, Tokyo
  - Research Site, Ome-shi, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Suginami-ku, Tokyo
  - Research Site, Tanabe-shi, Wakayama
  - Research Site, Wakayama, Wakayama
  - Research Site, Chuo-shi, Yamanashi
- South Korea (4):
  - Research Site, Cheonan, Chungcheongnam-do
  - Research Site, Daejeon
  - Research Site, Incheon
  - Research Site, Seoul
- Taiwan (4):
  - Research Site, Niao-song-shiang, Kaohsiung
  - Research Site, Kweishan Shiang, Taoyuan Hsien
  - Research Site, Taichung
  - Research Site, Taipei

REFERENCES:
- See also: CSR-D5130C00027.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=473&filename=CSR-D5130C00027.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 817 patients were enrolled from 3 countries (Japan, South Korea and Taiwan). Of the randomised patients, most patients were Japanese (723 [90.3%]). The first patient was enrolled on 28 February 2010 and the last patient completed the study on 31 July 2012.
Pre-assignment Details: In total, 801 patients (401 in the ticagrelor [AZD6140 90 mg bd] group and 400 patients in the clopidogrel [clopidogrel 75 mg od] group) were randomised to treatment. The reasons for not being randomised were "Incorrect enrolment before randomisation" and "Patient decision (withdrawal of consent)".
Groups:
- Ticagrelor (AZD6140): Ticagrelor (AZD6140) 90 mg bid
- Clopidogrel: Clopidogrel 75mg od
Period: Overall Study
Arm/Group | Ticagrelor (AZD6140) | Clopidogrel
Started | 401 | 400
Received Randomized Treatment | 387 | 380
Completed | 335 | 337
Not Completed | 66 | 63
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 65 | 63

BASELINE CHARACTERISTICS:
Population: One discontinued patient (due to withdrawal of consent) in Ticagrelor (AZD6140) group did not agree to disclose any data. Thus the number of baseline participants in Ticagrelor (AZD6140) group is 400 instead of 401 that is the number of participants who started the first period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor (AZD6140) | Clopidogrel | Total
Number analyzed (Participants) | 400 | 400 | 800
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (12) | 66 (11) | 67 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 93 | 188
  Male | 305 | 307 | 612
Race/Ethnicity, Customized [Number; unit: Participants]
  Chinese | 16 | 19 | 35
  Japanese | 361 | 360 | 721
  Korean | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Major Bleeding
Description: Time to first occurrence of any major bleeding event (adjudicated by an independent Clinical Endpoint Committee (ICEC)). 1-year event rate (%) estimated via Kaplan-Meier method.
Time Frame: Ongoing up to12 months
Population: Safety analysis set which includes all patients who received randomized treatment with available post-treatment safety data
Measure: Number; unit: Percent probability
Groups:
- Ticagrelor (AZD6140): Ticagrelor (AZD6140) 90mg bid
Arm/Group | Ticagrelor (AZD6140) | Clopidogrel
Number analyzed (Participants) | 387 | 380
Percent probability | 11.2 | 8.4
Statistical Analysis 1: Comparison: Ticagrelor (AZD6140) vs Clopidogrel; No formal statistical comparison; Test type: Superiority or Other; Regression, Cox — No P-value provided since the objective was not to perform formal statistical comparison; Analyzed based on proportional hazards model including treatment group only; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.94 to 2.53] — Ticagrelor/Placebo

2. Primary Outcome: Major Adverse Cardiac Events (MACE)
Description: Time to first occurrence of any event from the composite of death from vascular causes, Myocardial Infarction (MI) and stroke (adjudicated by an ICEC). 1-year event rate (%) estimated via Kaplan-Meier method.
Time Frame: Ongoing up to 12 months
Population: Full Analysis set which includes all randomized patients with available post-randomization efficacy data
Measure: Number; unit: Percent probability
Arm/Group | Ticagrelor (AZD6140) | Clopidogrel
Number analyzed (Participants) | 400 | 400
Percent probability | 10.2 | 8.1
Statistical Analysis 1: Comparison: Ticagrelor (AZD6140) vs Clopidogrel; No formal statistical comparison based on hypothesis test; Test type: Superiority or Other; Regression, Cox — No P-value provided since the objective was not to perform formal statistical comparison; Analyzed based on proportional hazards model including treatment group only; Hazard Ratio (HR) = 1.47, 95% CI 2-sided [0.88 to 2.44] — Ticagrelor/Placebo

3. Secondary Outcome: Major and Minor Bleeding
Description: Time to first occurrence of any major or minor bleeding event (adjudicated by an independent Clinical Endpoint Committee (ICEC)). 1-year event rate (%) estimated via Kaplan-Meier method.
Time Frame: Ongoing up to12 months
Population: as for outcome 1
Measure: Number; unit: Percent probability
Arm/Group | Ticagrelor (AZD6140) | Clopidogrel
Number analyzed (Participants) | 387 | 380
Percent probability | 26.8 | 16.2
Statistical Analysis 1: Comparison: Ticagrelor (AZD6140) vs Clopidogrel; No formal statistical comparison; Test type: Superiority or Other; Regression, Cox — No P-value provided since the objective was not to perform formal statistical comparison; Analyzed based on proportional hazards model including treatment group only; Hazard Ratio (HR) = 1.72, 95% CI 2-sided [1.23 to 2.40] — Ticagrelor/Placebo

4. Secondary Outcome: Composite of All-cause Mortality, MI or Stroke
Description: Time to first occurrence of any event from the composite of death from any causes, Myocardial Infarction (MI) and stroke (adjudicated by an ICEC). 1-year event rate (%) estimated via Kaplan-Meier method.
Time Frame: Ongoing up to 12 months
Population: Full Analysis set which includes all randomized patients with available post-randomization efficacy data
Measure: Number; unit: Percent probability
Arm/Group | Ticagrelor (AZD6140) | Clopidogrel
Number analyzed (Participants) | 400 | 400
Percent probability | 10.5 | 8.1
Statistical Analysis 1: Comparison: Ticagrelor (AZD6140) vs Clopidogrel; No formal statistical comparison based on hypothesis test; Test type: Superiority or Other; Regression, Cox — No P-value provided since the objective was not to perform formal statistical comparison; Analyzed based on proportional hazards model including treatment group only; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.91 to 2.50] — Ticagrelor/Placebo

ADVERSE EVENTS:
Time Frame: Approximately 6 months to 1 year.
Arm/Group | Ticagrelor (AZD6140) | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 92/387 | 112/380
Other Adverse Events (participants affected / at risk) | 327/387 | 337/380
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor (AZD6140) (N=387) | Clopidogrel (N=380)
Coronary artery stenosis (Cardiac disorders) | 36 | 47
Angina pectoris (Cardiac disorders) | 5 | 9
Angina unstable (Cardiac disorders) | 4 | 5
Myocardial ischaemia (Cardiac disorders) | 2 | 3
Acute myocardial infarction (Cardiac disorders) | 4 | 2
Ventricular fibrillation (Cardiac disorders) | 3 | 1
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
supraventricular tachycardia (Cardiac disorders) | 1 | 0
Postinfarction angina (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 0 | 1
coronary artery perforation (Cardiac disorders) | 0 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 11 | 10
Coronary artery restenosis (Injury, poisoning and procedural complications) | 6 | 8
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 1
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 2 | 1
patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Fat embolism (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebral infarction (Nervous system disorders) | 4 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Brain stem stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Herpes Zoster (Infections and infestations) | 1 | 2
Pyelonephritis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Thrombosis in device (General disorders) | 2 | 4
Device occlusion (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 1
Loose tooth (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Radicular cyst (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 2
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumber spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Anomalous arrangement of pancreaticobiliary duct (Congenital, familial and genetic disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.8% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor (AZD6140) (N=387) | Clopidogrel (N=380)
Constipation (Gastrointestinal disorders) | 59 | 55
Diarrhoea (Gastrointestinal disorders) | 26 | 23
Vomiting (Gastrointestinal disorders) | 21 | 27
Nausea (Gastrointestinal disorders) | 21 | 26
Abdominal discomfort (Gastrointestinal disorders) | 9 | 9
Abdominal pain upper (Gastrointestinal disorders) | 10 | 3
Dental Caries (Gastrointestinal disorders) | 3 | 8
Myocardial infarcion (Cardiac disorders) | 35 | 23
Angina pectoris (Cardiac disorders) | 16 | 22
Coronary artery stenosis (Cardiac disorders) | 14 | 17
Bradycardia (Cardiac disorders) | 11 | 8
Cardiac failure (Cardiac disorders) | 8 | 8
Ventricular tachycardia (Cardiac disorders) | 8 | 8
Ventricular extrasystoles (Cardiac disorders) | 7 | 6
Atrial fibrillation (Cardiac disorders) | 5 | 10
Nasopharyngitis (Infections and infestations) | 55 | 59
Urinary tract infection (Infections and infestations) | 10 | 5
Pneumonia (Infections and infestations) | 8 | 3
Pyrexia (General disorders) | 56 | 51
Non-cardiac chest pain (General disorders) | 8 | 1
Oedema peripheral (General disorders) | 8 | 12
Puncture site pain (General disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 46
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 10
Eczema (Skin and subcutaneous tissue disorders) | 16 | 9
Rash (Skin and subcutaneous tissue disorders) | 13 | 20
Blister (Skin and subcutaneous tissue disorders) | 8 | 8
Dermatitis contact (Skin and subcutaneous tissue disorders) | 7 | 5
Erythema (Skin and subcutaneous tissue disorders) | 6 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 11
Insomnia (Psychiatric disorders) | 58 | 49
Restlessness (Psychiatric disorders) | 14 | 3
Headache (Nervous system disorders) | 33 | 57
Dizziness (Nervous system disorders) | 22 | 18
Hypoaesthesia (Nervous system disorders) | 7 | 12
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 13 | 12
Contusion (Injury, poisoning and procedural complications) | 10 | 8
Procedural pain (Injury, poisoning and procedural complications) | 7 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Hypertension (Vascular disorders) | 23 | 27
Hypotension (Vascular disorders) | 9 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 12 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 10 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 10 | 9
Anaemia (Blood and lymphatic system disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No